CLINICAL TRIAL: NCT01061424
Title: A Community-Academic Partnership to Improve Asthma Management in Latino Children
Brief Title: The Community United to Challenge Asthma
Acronym: Project CURA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Molly A. Martin, MD, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21HL087769-01A1 (NIH)
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Asthma
Keywords: pediatric asthma
MeSH Terms: conditions — Asthma | interventions — Community Health Workers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- mailed information (Active Comparator): information on asthma is mailed to the home on the same schedule as the other arm
  Interventions: Behavioral: mailed information
- community health worker (Experimental): community health worker provides home visits for education
  Interventions: Behavioral: community health worker

INTERVENTIONS:
Behavioral: community health worker — community health worker provides home visits for education
  Arms: community health worker
Behavioral: mailed information — information on asthma is mailed to the home on the same schedule as the other arm
  Arms: mailed information

SUMMARY:
This study compares an asthma self-management intervention, delivered to the family and tailored to their needs and cultural beliefs, to standard asthma education in high-risk Puerto Rican children in elementary school. The primary outcomes are asthma medication adherence and trigger reduction.

ELIGIBILITY:
Inclusion Criteria:

* Puerto Rican
* In elementary school
* Diagnosed with asthma

Exclusion Criteria:

* Not in school
* Mild intermittent asthma
* Well controlled asthma

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
medication adherence | 1 year

SECONDARY OUTCOMES:
trigger reduction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Molly A Martin, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Martin MA, Mosnaim GS, Olson D, Swider S, Karavolos K, Rothschild S. Results from a community-based trial testing a community health worker asthma intervention in Puerto Rican youth in Chicago. J Asthma. 2015 Feb;52(1):59-70. doi: 10.3109/02770903.2014.950426. Epub 2014 Aug 27. PMID 25162304
- [Derived] Martin MA, Thomas AM, Mosnaim G, Greve M, Swider SM, Rothschild SK. Home asthma triggers: barriers to asthma control in Chicago Puerto Rican children. J Health Care Poor Underserved. 2013 May;24(2):813-27. doi: 10.1353/hpu.2013.0073. PMID 23728047
- [Derived] Martin MA, Olson D, Mosnaim G, Ortega D, Rothschild SK. Recruitment, asthma characteristics, and medication behaviors in Midwestern Puerto Rican youth: data from Project CURA. Ann Allergy Asthma Immunol. 2012 Aug;109(2):121-7. doi: 10.1016/j.anai.2012.06.005. Epub 2012 Jun 26. PMID 22840253